CLINICAL TRIAL: NCT01653977
Title: Impact of Early Goal-directed Fluid Therapy in Hypovolemic Patients Undergoing Emergency Surgery A Prospective, Randomised, Open Trial
Brief Title: Impact of Early Goal-directed Fluid Therapy in Hypovolemic Patients Undergoing Emergency Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recrutment difficulties
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pavlovic Gordana, MD, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NAC 09-044
Record Dates: First submitted 2012-07-18; First posted 2012-07-31 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Hypovolemic Shock; Trauma; Emergency; Surgery
Keywords: Hypovolemic shock; trauma; emergency; surgery; GDT; Picco
MeSH Terms: conditions — Shock; Wounds and Injuries; Emergencies | interventions — Standard of Care; Vasoconstrictor Agents; point 4 composite resin; Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONTROL (Active Comparator): In the CONTROL group, the administration of fluid (250-500ml crystalloids or colloids) and cardiovascular supportive drugs will be guided to maintain standard pressure-related parameters within a normal range: MAP > 65mmHg, HR < 90/min, CVP >8-12< cm H20, urinary output > 0.5 ml/kg/h. In line with the conventional approach, other physiological parameters will also be targeted: T° > 35.5°C, Sp02 > 95%, lactate < 2.5 mmol/L, normalisation of the BE. The maximal infused volume of hydroxyethyl starch (Voluven®) will be 33 ml/kg.
  Interventions: Other: CONTROL
- OPTIMIZED (Active Comparator): In the OPTIMIZED group, the central venous catheter and the 4-French artery catheter (femoral or humeral access site) will be connected to a dedicated haemodynamic monitor (Pulsiocath, PV2024L; Pulsion Medical Systems AG, Munich, Germany).
  The administration of fluid (250-500ml crystalloids or colloids) and cardiovascular supportive drugs will be guided by an algorithm taking into account standard parameters (HR, MAP, lactate, Hb), as well as static and dynamic volumetric parameters (SVI, CI, GEDVI, EVLWI, SVV, PPV, PVI).
  Interventions: Other: OPTIMIZED

INTERVENTIONS:
Other: CONTROL — In the CONTROL group, the administration of fluid (250-500ml crystalloids or colloids) and cardiovascular supportive drugs will be guided to maintain standard pressure-related parameters within a normal range: MAP > 65mmHg, HR < 90/min, CVP >8-12< cm H20, urinary output > 0.5 ml/kg/h. In line with the conventional approach, other physiological parameters will also be targeted: T° > 35.5°C, Sp02 > 95%, lactate < 2.5 mmol/L, normalisation of the BE. The maximal infused volume of hydroxyethyl starch (Voluven®) will be 33 ml/kg.
  Other Names: Standard care; trauma; fluide balance; Vasopressors
  Arms: CONTROL
Other: OPTIMIZED — In the OPTIMIZED group, the central venous catheter and the 4-French artery catheter (femoral or humeral access site) will be connected to a dedicated haemodynamic monitor (Pulsiocath, PV2024L; Pulsion Medical Systems AG, Munich, Germany).
  The administration of fluid (250-500ml crystalloids or colloids) and cardiovascular supportive drugs will be guided by an algorithm taking into account standard parameters (HR, MAP, lactate, Hb), as well as static and dynamic volumetric parameters (SVI, CI, GEDVI, EVLWI, SVV, PPV, PVI).
  Other Names: Goal-directed therapy; Picco; Fluide balance optimized; Vasopressor; CI
  Arms: OPTIMIZED

SUMMARY:
This study compares the safety and efficacy of GDTs using standard pressure-related parameters vs. dynamic hemodynamic indices associated with fluid compartment monitoring, in trauma patients requiring emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Severe hypovolemic condition°
* Need for emergent interventional procedure under general anesthesia with an expected duration > 120 min.

Exclusion Criteria:

* Patients responding to early fluid resuscitation (20ml/kg) who don't require a CVC
* Neurotrauma (Glasgow Coma Score < 12) and/ or medullar trauma
* Known pregnancy or diagnosed by US or Ct-scan (> 14 weeks)
* Sustained cardiac arrhythmia (see Logbook P8)
* Known or diagnosed severe cardiac valvular dysfunction (stenosis, insufficiency) (see Logbook P8)
* Known or diagnosed intracardiac shunt: interventricular or atrial defect (see Logbook P8)
* Burn injury > 10%
* Needed emergency thoracotomy or ABC resuscitation protocol
* Pre-existing severe liver dysfunction(Child-Pugh class C)
* Do-not-resuscitate order, died within 48h of admission
* Ultra-emergent surgery with no further diagnostic investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Delta lactate | From randomization, for the duration of surgery and up to transfer from the operating room to the ICU or recovery room, an expected average of 6 hours.
  The primary study endpoint will be the difference between the baseline arterial blood lactate at the time of randomization and the value of the arterial blood lactate at the time of transfer from the emergency operating room (∆ lactate).

SECONDARY OUTCOMES:
Cardiovascular complications: myocardial infarct or congestive heart failure | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcome and surrogate biomarkers (Troponin-I and pro-BNP: day 1-2-3) will be recorded by extracting this specific data from the electronic medical file, until discharge, death or up to 28 days, whichever comes first.
Cerebral complications: stroke | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcomes at day 1-2-3 will be recorded by extracting this specific data from the electronic medical file, and until discharge, death or up to 28 days, whichever comes first.
Pulmonary complications: ALI/ARDS, bronchopneumonia | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcomes at day 1-2-3 will be recorded by extracting this specific data from the electronic medical file, and until discharge, death or up to 28 days, whichever comes first.
Pulmonary complications: respiratory insufficiency necessitating re-intubation | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcomes at day 1-2-3 will be recorded by extracting this specific data from the electronic medical file, and until discharge, death or up to 28 days, whichever comes first.
Surgical complications: re-operation for bleeding or infection | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcomes at day 1-2-3 will be recorded by extracting this specific data from the electronic medical file, and until discharge, death or up to 28 days, whichever comes first.
Renal complications: infection, urosepsis or renal insufficiency | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcome and surrogate biomarkers (Riffle score, creatinine: day 1-2-3) will be recorded by extracting this specific data from the electronic medical file, until discharge, death or up to 28 days, whichever comes first.
Duration of post-operative mechanical ventilation: in hours | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcomes at day 1-2-3 will be recorded by extracting this specific data from the electronic medical file, and until discharge, death or up to 28 days, whichever comes first.
Total duration of ventilation : days | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
  Clinical outcomes (ventilation free days) will be recorded by extracting this specific data from the electronic medical file, and until discharge, death or up to 28 days, whichever comes first.
Length of stay in the ICU: in days | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
Length of stay in hospital: in days | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
Mortality | From randomization up to 28 days
SOFA score measurement | From randomization : day 1, day 2, day 3
Death | Day 1, day 2, day 3 after randomization until hospital discharge or up to 28 days or death, whichever comes first.
Number of unexpected ICU admission | From randomization up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Pavlovic, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux universitaires de Genève, Geneva, Canton of Geneva, Switzerland